CLINICAL TRIAL: NCT07271862
Title: A Novel Laparoscopic Apical Promontofixation Technique With Simultaneous Perineal Reconstruction for Patients With Symptomatic Pelvic Organ Prolapse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riga East Clinical University Hospital (Other Government)
Collaborators: Pauls Stradins Clinical University Hospital (Other); University of Latvia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-A/24
Record Dates: First submitted 2025-11-20; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Organ Prolapse (POP); Urinary Incontinence , Stress; Urinary Incontinence (UI); Female Sexual Dysfunction (FSD); Quality of Life
Keywords: Pelvic organ prolapse; Stress urinary incontinence; Urinary incontinence.; Female sexual dysfunction; Laparoscopic sacropexy; Mesh associated complications
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical technique (Active Comparator): Laparoscopic sacrocolpopexy.
  Interventions: Procedure: Laparoscopic sacrocolpopexy.
- Modified technique (Sham Comparator): Laparoscopic apical promontofixation combined with simultaneous vaginal and perineal reconstruction using native tissues.
  Interventions: Procedure: Laparoscopic apical promontofixation combined with simultaneous vaginal and perineal reconstruction using native tissues.

INTERVENTIONS:
Procedure: Laparoscopic sacrocolpopexy. — Laparoscopic sacrocolpopexy using a polypropylene mesh implant fixed to the cervix and along the entire anterior vaginal wall up to the bladder neck, with additional fixation along the posterior vaginal wall and to the levator ani muscles, ensuring physiological tension by securing the implant proximally to the sacral promontory, precisely to the anterior longitudinal vertebral ligament. Separate intracorporeal nonabsorbable sutures will be placed 1.5-2.0 cm apart. The following parameters will be analyzed: frequency and severity of intraoperative and postoperative complications (early and late), duration of surgery, length of hospital stay, recurrence rate, sexual activity, quality of life before and after surgery, as well as anatomical and functional outcomes. Anatomical results will be evaluated according to the POP-Q classification. Functional outcomes will be assessed using standardized questionnaires, including PFDI-20, FSFI, ICIQ in addition to urodynamic testing.
  Arms: Classical technique
Procedure: Laparoscopic apical promontofixation combined with simultaneous vaginal and perineal reconstruction using native tissues. — The procedure includes placement of a polypropylene implant with distal fixation to the bilateral uterosacral ligaments (according to the McCall technique) and to the cervix, as well as along the anterior vaginal wall up to the bladder neck, maintaining physiological tension, with proximal fixation to the sacral promontory, precisely to the anterior longitudinal vertebral ligament. A simultaneous colpoperineolevatoroplasty will also be performed. During the laparoscopic stage, separate intracorporeal nonabsorbable sutures will be placed 1.5-2.0 cm apart. During the vaginal stage, posterior colporrhaphy with simultaneous levatoroplasty for rectocele repair will be performed in patients with posterior vaginal wall prolapse or perineal defects. Parameters will be analyzed: frequency of intraoperative and postoperative complications, duration of surgery, length of hospital stay, sexual activity, quality of life before and after surgery, as well as anatomical and functional results.
  Arms: Modified technique

SUMMARY:
Pelvic organ prolapse in women is a common gynecological condition worldwide, with prevalence reported by different authors ranging from 15% to 50%. Up to 20% of women require surgical intervention during their lifetime due to genital prolapse or urinary incontinence. Surgical correction of prolapse provides an immediate effect by restoring the anatomical and physiological position of the pelvic organs, while also improving women's daily quality of life. Approximately 80-90% of women report satisfaction with the outcomes of prolapse surgery. However, there is still no global consensus regarding the optimal technique for performing colposacropexy. Multiple surgical approaches are currently in use, which prevents a definitive evaluation of the best method for surgical management of this condition. The classical laparoscopic sacrocolpopexy technique, while effective, does not eliminate the risk of mesh-related complications, particularly when synthetic implants are placed along the full length of the anterior and posterior vaginal walls.

Therefore, there is a strong rationale for developing a novel, simplified surgical approach for prolapse correction, derived from the original laparoscopic apical promontofixation, with simultaneous correction of cystocele and rectocele. This could potentially improve surgical outcomes for patients with pelvic organ prolapse while reducing the risk of complications associated with synthetic mesh implantation.

DETAILED DESCRIPTION:
This is a prospective randomized study conducted at Riga East University Hospital (Latvia) and Pauls Stradins Clinical University Hospital (Latvia). Two groups of female patients will be compared. In the first group, patients will undergo laparoscopic reconstructive pelvic organ prolapse surgery using a polypropylene implant according to the 'classical' technique, involving fixation to the levator ani muscle and promontofixation. In the second group, patients will undergo a novel laparoscopic reconstructive pelvic organ prolapse procedure using a polypropylene implant based on a 'modified' technique, consisting of laparoscopic apical promontofixation combined with vaginal and perineal tissue repair using native tissues.

Group1 (Classical technique): Half of the patients will undergo laparoscopic sacrocolpopexy using a polypropylene mesh implant fixed to the cervix and along the entire anterior vaginal wall up to the bladder neck, with additional fixation along the posterior vaginal wall and to the levator ani muscles, ensuring physiological tension by securing the implant proximally to the sacral promontory, precisely to the anterior longitudinal vertebral ligament. Separate intracorporeal nonabsorbable sutures will be placed 1.5-2.0 cm apart.

Group2 (Modified technique): Half of the patients will undergo laparoscopic apical promontofixation combined with simultaneous vaginal and perineal reconstruction using native tissues. The procedure includes placement of a polypropylene implant with distal fixation to the bilateral uterosacral ligaments (according to the MacCall technique) and to the cervix, as well as along the anterior vaginal wall up to the bladder neck, maintaining physiological tension, with proximal fixation to the sacral promontory, precisely to the anterior longitudinal vertebral ligament. A simultaneous colpoperineolevatoroplasty will also be performed. During the laparoscopic stage, separate intracorporeal nonabsorbable sutures will be placed 1.5-2.0 cm apart. During the vaginal stage, posterior colporrhaphy with simultaneous levatoroplasty for rectocele repair will be performed in patients with posterior vaginal wall prolapse or perineal defects.

The following parameters will be analyzed: frequency and severity of intraoperative and postoperative complications (early and late), duration of surgery, length of hospital stay, recurrence rate, sexual activity, quality of life before and after surgery, as well as anatomical and functional outcomes. Anatomical results will be evaluated according to the Pelvic Organ Prolapse Quantification System classification. Functional outcomes will be assessed using standardized questionnaires, including Pelvic Floor Distress Inventory-20, Female Sexual Function Index, and International Consultation on Incontinence Questionnaire, in addition to urodynamic testing. Anatomical and functional results, quality of life, and sexual activity will be analyzed over a 6-month postoperative follow-up period.

Based on the study results, the novel laparoscopic apical promontofixation technique with simultaneous perineal repair using native tissues will be introduced into clinical practice in hospitals providing gynecological care. Furthermore, a new unified clinical protocol will be developed to facilitate practical application, including a simplified diagnostic algorithm based on 4-6 key symptoms, enabling family physicians and outpatient gynecologists to identify women with pelvic organ prolapse and refer them for specialist evaluation and appropriate treatment planning.

Additionally, a new objective method for assessing the degree of prolapse will be developed, allowing specialists to more accurately measure anterior, posterior, and central vaginal wall defects. This method will involve specific markings on a gynecological plastic speculum, enabling more precise evaluation of vaginal wall defects during routine gynecological examination. The new method will also be compared with other internationally recognized approaches for surgical management of pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with symptomatic isolated or combined forms of pelvic organ prolapse, corresponding to stage II-IV according to the POP-Q classification.
2. Age between 30 and 80 years.
3. Presence or absence of urinary incontinence symptoms.
4. Preoperatively verified by urodynamics: occult, mild, or severe stress urinary incontinence, or absence thereof.
5. Presence or absence of proctogenic constipation.
6. No prior surgical interventions for pelvic organ prolapse or urinary incontinence.
7. History of supracervical hysterectomy.

Exclusion Criteria:

1. Severe extragenital pathology contraindicating surgical treatment.
2. Malignant pelvic pathology.
3. Asymptomatic patients.
4. Patient refusal to undergo subtotal hysterectomy.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-10-04 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Anatomical success after pelvic organ prolapse surgery. | Before and 6 months after surgery.
  Anatomical outcome will be assessed using the Pelvic Organ Prolapse Quantification (POP-Q) system. Success is defined as no prolapse beyond the hymen in any vaginal compartment. Unit of Measure: POP-Q stage (0-4).

SECONDARY OUTCOMES:
Functional outcome - pelvic floor symptoms. | Before and 6 months after surgery.
  Evaluation with standardized questionnaires: Pelvic Floor Distress Inventory (PFDI-20). Unit of Measure: PFDI-20 score (0-300).
Sexual function. | Before and 6 months after surgery.
  Female Sexual Function Index (FSFI) questionnaire to assess sexual activity and satisfaction. Unit of Measure: FSFI score (2-36).
Urinary function. | Before and 6 months after surgery.
  International Consultation on Incontinence Questionnaire (ICIQ) and urodynamic testing. Unit of Measure: ICIQ score (0-21); presence/absence of urodynamic abnormalities.
Postoperative complications. | Early (within 30 days) and late (up to 6 months) after surgery.
  Frequency and severity of intraoperative and postoperative complications (classified according to Clavien-Dindo). Unit of Measure: Number of events and severity grade.
Operative time. | 3 hours.
  Intraoperative.
Length of hospital stay. | 7 Days.
  From surgery until discharge.

OTHER OUTCOMES:
Quality of life. | Before and 6 months after surgery.
  Assessed using validated patient-reported outcome measures (PFDI-20 global score, condition-specific questionnaires). Unit of Measure: Questionnaire scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Riga East Clinical University Hospital. Pauls Stradins Clinical University Hospital., Riga, Latvia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol